CLINICAL TRIAL: NCT07089628
Title: Investigation of the Relationship Between Core Stability and Reaction Time, Hand-Eye Coordination, Pain, and Functional Status in Individuals With Rotator Cuff Lesions
Status: Recruiting | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Eren Ozen, Principal Investigator, Bandırma Onyedi Eylül University
Other Study IDs: 2025 - 985
Record Dates: First submitted 2025-07-21; First posted 2025-07-28 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Core Stability; Core Stabilization; Reaction Time; Pain; Function
Keywords: Core Stability; Core Stabilization; Reaction time; Hand- Eye Coordination; Pain; Function
MeSH Terms: conditions — Pain | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rotator Cuff Lesion Group: This group will consist of individuals with rotator cuff lesions. The assessments described will be conducted on these participants.
  Interventions: Other: Assessment
- Control Group: This group will include asymptomatic control participants, consisting of patient relatives, university staff, and students who have no shoulder problems and are matched in terms of age, sex, and educational level.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — There is no intervention in this study. Participants will only undergo assessments.

SUMMARY:
Rotator cuff lesions are among the most common problems within musculoskeletal disorders. The prevalence of these lesions increases with age, and they encompass a wide spectrum of various injuries and pathological conditions. The literature frequently reports that such lesions often lead to pain, decreased functional capacity, and a reduction in quality of life. Although some of these lesions are traumatic in origin, the majority of rotator cuff problems are degenerative due to age-related changes in tendon structure.

Recent scientific studies have indicated that core stability may be a significant factor in such musculoskeletal problems. Adequate core stabilization not only minimizes the load on the vertebral column but also enhances the strength and endurance of peripheral joints and facilitates the transfer of energy to distal segments. Given that rotator cuff lesions can adversely affect upper extremity functions and potentially result in reduced core stability, we hypothesize that they may negatively influence reaction time and hand-eye coordination, which are essential for the effective execution of motor tasks.

To date, no studies have been identified in the literature investigating the relationship between core stability and reaction time or hand-eye coordination in individuals with rotator cuff lesions. In light of this information, the aim of our planned study is to examine the relationship between core stability and reaction time, hand-eye coordination, pain, and functional status in individuals with rotator cuff lesions and to compare these findings with asymptomatic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of a rotator cuff lesion confirmed by a physician
* Having no history of any surgical procedure related to the shoulder
* Experiencing activity-related pain scored as 3 or higher on the Visual Analog Scale

Exclusion Criteria:

* Presence of systemic inflammatory diseases
* Pregnancy
* Presence of mental health disorders
* Individuals with communication difficulties
* Presence of other significant shoulder pathologies such as dislocation, fracture, arthritis, or frozen shoulder

  * All of these criteria apply to the group with rotator cuff lesions. The other group consists of healthy, asymptomatic individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: "Rotator cuff lesions are among the most common problems within musculoskeletal disorders. The prevalence of these lesions increases with age, and they encompass a wide spectrum of various injuries and pathological conditions. The literature frequently reports that these lesions often result in pain, reduced functional capacity, and a decline in quality of life. Although some of these lesions are traumatic in nature, the majority of rotator cuff issues are degenerative due to age-related changes in tendon structure.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified "Biering-Sorensen" test | Baseline
  Test will be applied to assess the endurance of the core muscles. The subjects are positioned in the prone position. The subjects are asked to extend their upper body straight forward from the edge of the table. How long the patient was able to perform the test was recorded in seconds.
Trunk flexors endurance test | Baseline
  Test will be applied to assess the endurance of the core muscles. Participants will be positioned with trunk flexed to 60º, knees and hips to 90º flexion. The evaluator fixes the feet on the ground by supporting them from the toes. When the 60º trunk flexion is broken, the test will be terminated. How long the patient was able to perform the test was recorded in seconds.
Lateral bridge test | Baseline
  Test will be applied to assess the endurance of the core muscles. The subjects were asked to lie on their side, raise their bodies on their forearms and toes and maintain this position(both sides). How long the patient was able to perform the test was recorded in seconds.
Prone bridge test | Baseline
  Test will be applied to assess the endurance of the core muscles. The subjects put their elbows on the ground as the starting position and open their feet about the width of their hips while keeping their body straight. The tests end when the subjects break the test positions. How long the patient was able to perform the test was recorded in seconds.
Modified "Push-ups" test | Baseline
  Test will be applied to assess the strength of the core muscles. The subjects are positioned in the prone position with their hands shoulder-width apart and elbows and knees flexed. The subjects were asked to raise their body up by extending their elbows. The number of times the patient repeats the movement in 30 seconds is recorded.
Sit-ups test | Baseline
  Test will be applied to assess the strength of the core muscles. The subjects are asked to flex the trunk while the knees are flexed in the supine position. During the test, the feet of subjects are stabilized. The number of times the patient repeats the movement in 30 seconds is recorded.

SECONDARY OUTCOMES:
Reaction Time | Baseline
  In this study, the BlazePod system will be used to measure reaction time. BlazePod is a mobile application-supported system that records response time to visual stimuli with millisecond precision through LED light pods. Prior to the assessment, a pre-test will be conducted to allow participants to adapt to the evaluation process. The right and left sides will be assessed separately. During a 30-second period, the number of extinguished LEDs, the average time to deactivate each LED (in milliseconds), and the number of missed LEDs-defined as those that automatically turn off after the designated waiting period-will be recorded.
Hand-Wall Toss Test | Baseline
  Hand-eye coordination will be assessed using the Hand-Wall Toss Test. During the test, participants will be instructed to stand 2 meters away from the wall and throw a tennis ball at the wall with their right hand, catching it with their left hand, and then alternate hands, continuing this sequence for 30 seconds. The total number of successful wall tosses and catches performed without dropping the ball will be recorded.
Visual Analogue Scale | Baseline
  It is used to assess the severity of pain. Pain severity with Visual Analogue Scale,(0-10) higher scores indicate more pain.
Shoulder Pain and Disability Index | Baseline
  Shoulder function will be assessed using the Shoulder Pain and Disability Index (SPADI). The SPADI consists of two sections-pain and disability-with a total of 13 items. Each item is scored on a scale from 0 to 10, and the results are calculated as a percentage. The total score ranges from 0 to 100, with higher scores indicating worse shoulder functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Hazar, Prof., Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)